CLINICAL TRIAL: NCT02676908
Title: A Randomised Controlled Trial Comparing Duration of Compression Hosiery After Endovenous Ablation of Varicose Veins
Brief Title: Optimum Duration of Compression Stockings After Endovenous Varicose Vein Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Caitriona Canning, Fellow in Vascular Medicine, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJH-01-VV
Record Dates: First submitted 2015-08-06; First posted 2016-02-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Varicose Veins
Keywords: endovenous ablation; laser; radiofrequency; stockings
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4 weeks & EVLT (No Intervention): After endovenous laser therapy and avulsions, patients will wear compression socks for four weeks (usual care)
- 4 weeks & RFA (No Intervention): After radiofrequency ablation therapy and avulsions, patients will wear compression socks for four weeks (usual care)
- 2 weeks & EVLT (Experimental): After endovenous laser therapy and avulsions, patients will wear compression socks for two weeks (trial group)
  Interventions: Other: Compression socks for 2 weeks
- 2 weeks & RFA (Experimental): After radiofrequency ablation therapy and avulsions, patients will wear compression socks for two weeks (trial group)
  Interventions: Other: Compression socks for 2 weeks

INTERVENTIONS:
Other: Compression socks for 2 weeks — Patients in the intervention group will be asked to wear compression stockings for two weeks post-operatively
  Arms: 2 weeks & EVLT; 2 weeks & RFA

SUMMARY:
Compression stockings are traditionally worn for a period of time after varicose vein surgery to reduce pain and bruising. The investigators provide an ambulatory endovenous ablation service. Patients come to the Veins Unit, receive oral sedation, have their veins treated with either laser or radiofrequency ablation plus phlebectomies* under local anaesthetic, recover for an hour and then go home. *Phlebectomy describes the technique of pulling out small varicose veins through small incisions in the overlying skin. The standard practice of the Veins Unit is to advise patients to wear class two compression stockings for four weeks post-operatively. Many patients would prefer a shorter period of time in stockings.

The Nice Guidelines for Varicose Veins has posed the question: 'How long should stockings be worn for after endovenous ablation?'

Three trials have addressed this issue:

Bakker looked at patients who wore stockings for either two or seven days after laser ablation only; the group who wore stockings for seven days fared better.

Elderman looked at patients who either wore no stockings or stockings for two weeks after laser ablation only; the group who wore stockings for two weeks had less pain.

Krasznai looked at patients who wore stockings for either 4 hours or 72 hours after radiofrequency ablation only; there was no significant difference in post-op pain among groups.

None of these trials included patients who had phlebectomies at the same time. This study aims to answer the question 'How long is it necessary to wear compression stockings for after endovenous ablation (either laser or radiofrequency) plus concomitant phlebectomies?' The investigators plan to divide 110 patients into two groups- either 'stockings for 2 weeks' (trial group) or 'stockings for 4 weeks' (usual treatment group).

Pre-operatively, all patients will fill out a pain score and two short quality of life questionnaires, one specific to varicose veins. Post-operatively at home, all patients will be asked to keep a diary of pain and analgesia use. They will also document bruising at seven days on charts and on a visual scale. At their four week clinic review, all patients will be asked to fill out a pain and bruising score, a bruising chart and the two short quality of life questionnaires again.

The group with the best pain, bruising and quality of life scores post-operatively will help guide duration of compression therapy for future patients.

DETAILED DESCRIPTION:
The Nice Guidelines for Varicose Veins, published by the NHS in 2013, questioned the clinical benefit of stockings after endovenous ablation, and if there is benefit, how long the stockings should be worn for.

Three randomised controlled trials have addressed these issues:

Bakker and colleagues randomised 69 patients into two groups- stockings were worn for either two or seven days after laser ablation. The group who wore stockings for seven days had better pain and quality of life scores.

Elderman and colleagues randomised 111 patients who had laser ablation into two groups- a group who wore no stockings, or a group who wore stockings for two weeks. The group who wore stockings for two weeks had less pain and required less analgesia.

Krasznai and colleagues randomised 101 patients into two groups- stockings were worn for either 4 hours or 72 hours after radiofrequency ablation only; there was no significant difference in post-op pain among groups.

None of these trials included patients who had phlebectomies at the same time.

This study hopes to answer the question 'How long is it necessary to wear compression stockings for after endovenous ablation (either laser or radiofrequency) plus concomitant phlebectomies?'

110 consecutive patients will be randomised into 'stockings for 2 weeks' (trial group) or 'stockings for 4 weeks' (usual treatment group). Randomisation will be facilitated by online random number generation (https://www.random.org/). Patients with odd numbers will be allocated into the trial group; those randomly assigned even numbers will be allocated into the usual treatment group.

Pre-operatively, all patients will be asked to fill out a visual analog pain score (VAS), the Aberdeen Varicose Veins questionnaire and the RAND 36-Item Health Survey. Patients will be evaluated in terms of CAEP staging and the Venous Clinical Severity Score (VCSS) by the supervising nurse or physician.

Endovenous laser therapy (EVLT) plus phlebectomies or radiofrequency ablation (RFA) plus phlebectomies will be performed in the standard manner.

The trial group will wear the stockings for 24 hours a day for the first 4 days, and then during the day only for the next 10 days. The usual treatment group will wear the stockings for 24 hours a day for a week, and then during the day only for the next 3 weeks.

Post-operatively at home, patients will be asked to keep a diary of pain and analgesia use. They will also document bruising at 7 days on a diagram and on a visual analog scale.

At their 4 week clinic review, again the VCSS will completed and patients will be asked to fill out a visual analog pain and bruising score, a bruising diagram, the Aberdeen Varicose Veins questionnaire and the RAND 36-Item Health Survey.

Primary outcome measures are post-operative pain scores on the visual analog scale and post-operative bruising scores on the visual analog scale.

Secondary outcome measures are changes in veins-related quality of life measured on the Aberdeen Varicose Veins Questionnaire and changes in overall quality of life based on the RAND 36-Item Health Survey.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent varicose veins
* Diagnosis on duplex of truncal (GSV and/or SSV and/or AATV) insufficiency
* Must be able to provide informed consent

Exclusion Criteria:

* Patients who require long term compression (active ulcers/ deep venous incompetence)
* Patients who have already had one leg enrolled in the study
* Patients with congenital venous malformations
* Patients who require avulsions only
* Patients who are unable to complete the questionnaires due to a lack of command over the language or who have vision/ hearing disabilities
* Patients who are unable to attend the hospital for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | Change from baseline at four weeks

SECONDARY OUTCOMES:
Quality of Life (Veins Related) | Change from baseline at four weeks
  Changes in veins related quality of life based on the Aberdeen Varicose Veins Questionnaire
Quality of Life (General) | Change from baseline at four weeks
  Changes in general quality of life based on the RAND 36-Item Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- St James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker NA, Schieven LW, Bruins RM, van den Berg M, Hissink RJ. Compression stockings after endovenous laser ablation of the great saphenous vein: a prospective randomized controlled trial. Eur J Vasc Endovasc Surg. 2013 Nov;46(5):588-92. doi: 10.1016/j.ejvs.2013.08.001. Epub 2013 Sep 5. PMID 24012465
- [Background] Krasznai AG, Sigterman TA, Troquay S, Houtermans-Auckel JP, Snoeijs M, Rensma HG, Sikkink C, Bouwman LH. A randomised controlled trial comparing compression therapy after radiofrequency ablation for primary great saphenous vein incompetence. Phlebology. 2016 Mar;31(2):118-24. doi: 10.1177/0268355514568658. Epub 2015 Jan 23. PMID 25616874
- See also: Elderman JH, Krasznai AG, Voogd AC, Hulsewé KWE, Sikkink CJJM. Role of compression stockings after endovenous laser therapy for primary varicosis. JVS Venous and Lymphatic Disorders. 2014 2(3): 289-296 — http://dx.doi.org/10.1016/j.jvsv.2014.01.003